CLINICAL TRIAL: NCT00088296
Title: Effects of Osteoarthritis Pain, Morphine and Placebo on Neuro-Endocrine Function in Men
Brief Title: Effects of Osteoarthritis Pain, Morphine, and Placebo on Neuroendocrine Function in Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040239; 04-AT-0239
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-18

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; MS Contin; Placebo; Cortisol; Testosterone; Degenerative Joint Disease; OA; Arthritis; Joint Pain; Arthritic Pain; Opioid
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Arthritis; Arthralgia | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood Draw

SUMMARY:
This study will examine the effects of morphine on leuteinizing hormone, testosterone, adrenocorticotropic hormone and cortisol in men. The use of long-term opioids, such as morphine, to treat patients with pain is increasing, despite a dearth of information about their effects on hormones. The study will also look at the effect of chronic pain on these hormone levels and the effect of placebo on pain.

Men between 30 and 65 years of age who have had moderate to severe chronic pain due to osteoarthritis for at least 3 months and healthy, pain-free men in the same age range may be eligible for this study. Patients taking an opioid-based medication such as percocet, vicodin, or morphine for pain relief, as well as patients who are not taking opioids, may participate. Candidates are screened with a medical history, physical examination, blood tests, including a blood test to look for possible "pain genes," electrocardiogram, x-ray, and questionnaires that assess the impact of pain on functional level and psychological well being.

This is a four-part study. Healthy volunteers and patients who are taking opioids for their arthritis pain end their participation after Part I; those who are not taking opioids continue with Parts II, III, and IV, as follows:

Part I: Participants are admitted to the NIH Clinical Center at 4 p.m. for an overnight stay. At 6 p.m. a catheter (plastic tube) is placed in a vein in the forearm and remains in place throughout the night. Blood samples of 3 cc's each (less than a teaspoon) are collected through the catheter every 20 minutes for 12 hours, from 8 p.m. until 8 a.m. Participants also collect their urine starting from 8 a.m. on the morning of hospital admission and continue the collection throughout their 24-hour hospital stay. Patients are discharged at the completion of the blood sampling.

Part II: Patients are randomly assigned to take morphine (MS Contin), placebo, or standard treatment, which consists of anti-inflammatory medications and acetaminophen as needed, but no opioids. (Patients in groups I and II are also permitted to take anti-inflammatory drugs and acetominophen, in addition to their study medication.) Patients are monitored for drug side effects by phone twice a week, and medication doses are adjusted as needed. The morphine dose is gradually increased over a 4-week period if no side effects develop. After 2 weeks on the highest dose of morphine, hormone blood levels are measured and patients complete questionnaires. Patients are readmitted to the hospital for a repeat blood sampling and blood collection as in Part I. Patients on morphine and placebo are then gradually tapered off drug over 12 days and remain drug-free for 2 days before starting Part III.

Part III: All patients are given morphine in this part of the study and are monitored for drug side effects by phone twice a week, with doses adjusted as needed. The morphine is gradually increased over a 6-week period if no side effects develop and is maintained at the highest dose for another 8 weeks. Hormone levels are measured and the blood and urine studies and questionnaires are repeated. Patients interested in continuing long-term treatment with MC Contin are referred back to their physicians with recommendations to that effect.

Part IV: Patients are followed by phone for 6 months, at which time they return to the Clinical Center for hormone level measurements, repeat blood and urine tests, and questionnaires.

DETAILED DESCRIPTION:
Several studies suggest that acceptance and use of opioid medicines for relief of chronic pain are increasing substantially, and that opiodergic medications and chronic pain each perturb neuroendocrine functions, especially those of the hypothalamic pituitary, adrenal, and gonadal axes. The objectives of the proposed protocol, entitled "Effects of Chronic Musculoskeletal Pain and Opioidergic versus Placebo Interventions on Neuro-endocrine Function in Men," are three fold:

1. To determine whether long term opioid usage in men with chronic pain due to osteoarthritis results in abnormalities of ACTH, cortisol, LH and testosterone secretion.
2. To evaluate whether placebo analgesia results in a similar hormonal response as elicited by an opioid analgesic. Prior imaging studies have shown that placebo analgesia is associated with activation of similar parts of the cortex as with analgesic intake.
3. To evaluate the effects of chronic pain per se on ACTH, cortisol, LH and testosterone secretion.

To address these questions, we propose a 4-part study. In part I, 12 healthy men will be compared with 12 men with chronic osteoarthritis (OA) pain on long term opioids and 12 narcotic naive men with chronic OA pain by means of 12 hour overnight frequent blood sampling for measurement of cortisol, ACTH, LH and testosterone.

In part II, 36 narcotic naive patients with chronic OA, pain, all of whom will have undergone overnight hormone sampling in Part I, will be randomized to one of three treatment groups: MS Contin (15-90 mg), placebo and "standard treatment."

Doses of placebo and MS Contin will be escalated over 4 weeks in a similar fashion with two-week maintenance and 2 week taper. At the end of maintenance at 6 weeks, all patients will return for repeat 12 hour frequent sampling of the same hormones as in Part I. At the end of part II, patients will be invited to go on to an open label treatment period with MS Contin (15-120 mg) in part III of the study, which will consist of 6-week dose escalation and 8 weeks maintenance. At that point patients will be referred back to their physicians with recommendations for continued treatment with MS Contin, if patients are interested in this option.

Patients will be followed by phone for 6 months. At that point they will be asked to return to clinic for part IV, an outpatient AM sample of testosterone, LH, ACTH and cortisol. The primary endpoints of this study will be measures of LH, testosterone, ACTH, and cortisol secretion, whereas the secondary endpoints will be neurobehavioral indices such as pain and bothersomeness on visual analog scales, the Oswestry Disability Index, Multidimensional Pain Inventory, and the Beck Depression Inventory. It is anticipated that this study will provide novel information regarding the effects of chronic musculoskeletal pain, and treatment with opioids versus placebo, on selected neuroendocrine functions in men.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Clinical evidence of chronic OA by history and examination in a major joint or the spine.

     1. Pain level of 4/10 or greater on a scale of 0 to 10
     2. Pain for a duration of 3 months or longer present at least 5 out of 7 days a week
     3. Radiographic evidence of moderate to severe OA in the involved joint based on the Kellgren and Lawrence scoring scale.
  2. Age between 30-65 at study entry
  3. Men of all ethnicities
  4. Ability to understand the study measures and mentally capable of giving consent to participate in the study (based on an 8th grade education level)
  5. Willingness to refrain from taking opioids other than as dictated by the study design

EXCLUSION CRITERIA :

1. Impaired pulmonary, renal, hepatic, cardiovascular or endocrine-metabolic function; major coexisting medical condition such as cancer, chronic obstructive pulmonary disease and severe hepatic and renal dysfunction
2. Primary or secondary endocrine disease such as diabetes or Cushing's syndrome
3. Prostatic disease requiring usage of urological medications
4. Presence of sexual dysfunction defined as lack of libido, impotence or erectile abnormalities.
5. Current symptoms of coronary artery disease
6. Presence of RA, or other types of inflammatory arthritis
7. Use of systemic corticosteroids in the two months before screening and study entry
8. Alcohol abuse up to a year prior to study enrollment
9. Usage of any recreational drugs
10. History of narcotic abuse at any time in the past
11. Major depression whether successfully or unsuccessfully treated or diagnosed at the time of study screening based on a score of greater than or equal to 20 on the Beck Depression Inventory
12. Hct less than 35; anemia or bleeding disorder
13. Allergy to morphine
14. Current or past history of fibromyalgia as described by Wolfe F et al., (1990) (a minimum of 12 out of 19 points of tenderness must be present to satisfy criteria for fibromyalgia)
15. Cognitive impairment such that the individual is unable to give informed consent, complete study data collection tools or required study visits
16. Age 29 years or less due to rarity of OA in this age group
17. Body mass index (BMI) greater than 30kg/m(2) and BMI less than 20kg/m(2)

Usage of nonsteroidal anti-inflammatory drugs (NSAIDs) will be allowed at study entry and during the conduct of the study. Patients will be asked to refrain from using muscle relaxers, other opioids apart from the study drug (MS Contin), AED's (anti-epileptic drugs), TCAs (tricyclic antidepressants), SSRIs (selective serotonin reuptake inhibitors) and benzodiazepines for pain control during part II and III. Patients will also be asked to refrain from having local joint injections with steroids or other agents. Patients will be queried regarding their use of complementary and/or alternative medicine (CAM) treatments (e.g. acupuncture, chiropractic manipulations, herbs and botanicals, and mind-body interventions) at the start of the study and will be counseled against beginning CAM treatments during the study protocol. Starting any of these treatments during the study will be considered a study violation. The only exception will be for glucosamine and/or chondroitin.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-07-13; Study Completion 2007-10-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Celani MF, Carani C, Montanini V, Baraghini GF, Zini D, Simoni M, Ferretti C, Marrama P. Further studies on the effects of heroin addiction on the hypothalamic-pituitary-gonadal function in man. Pharmacol Res Commun. 1984 Dec;16(12):1193-203. doi: 10.1016/s0031-6989(84)80084-3. PMID 6522443